CLINICAL TRIAL: NCT05214911
Title: Multicenter,Randomized, Parallel,Double-blind, Comparative Study of the Superiority of the Desloratadine 0.5mg/mL and Prednisolone 4 mg/mL Versus Desloratadine 0.5mg/mL in the Treatment of Persistent Allergic Rhinitis in Children (DESPRED)
Brief Title: Fixed Dose Combination of Desloratadine / Prednisolone in the Treatment of Moderate Severe Allergic Rhinitis in Children
Acronym: DESPRED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EF177
Record Dates: First submitted 2021-12-13; First posted 2022-01-31 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — desloratadine; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind, double-dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental drug (Desloratadine 0.5 mg/mL/Prednisolone 4 mg/mL) (Experimental): ADF Group 1 - Eurofarma drug association of Desloratadine 0.5 mg/mL / Prednisolone 4 mg/mL
  Interventions: Drug: Desloratadine , Prednisolone
- Active Comparator: Desalex® (Desloratadine 0.5 mg/mL) (Active Comparator): Desalex® Group 2 - Eurofarma drug Desloratadine 0.5 mg/mL
  Interventions: Drug: Desloratadine

INTERVENTIONS:
Drug: Desloratadine , Prednisolone — FDC desloratadine 0.5 mg/mL/prednisolone 4 mg/mL from Eurofarma Laboratórios SA
  Arms: Experimental drug (Desloratadine 0.5 mg/mL/Prednisolone 4 mg/mL)
Drug: Desloratadine — Desloratadine 0.5 mg/mL (Desalex® - Eurofarma Laboratórios SA)
  Arms: Active Comparator: Desalex® (Desloratadine 0.5 mg/mL)

SUMMARY:
Multicenter, randomized, parallel-group, double-blind, double-dummy, comparative clinical trial of the superiority of the fixed-dose combination of desloratadine 0.5 mg/mL and prednisolone 4 mg/mL from Eurofarma Laboratórios SA versus desloratadine 0.5 mg/mL in the treatment of moderate to severe persistent allergic rhinitis in children aged 6 to 12 years.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

DETAILED DESCRIPTION:
Desloratadine and prednisolone are active pharmaceutical ingredients (APIs) already registered in the country as monodrugs. These products are widely used and their efficacy and safety are well known in daily clinical practice in the approved indications.

Once confirmed the absence of pharmacokinetic interaction between desloratadine and prednisolone in relative bioavailability studies, this phase 3 study will be conducted with the objective of demonstrating the superiority of the new FDC containing desloratadine and prednisolone over the isolated administration of desloratadine in treatment from moderate to severe allergic rhinitis in children. The aim is to provide a new effective, safe and well-tolerated therapeutic option for dealing with these cases.

Multicenter, randomized, parallel group, double blind, double-dummy, superiority comparative clinical trial.

Children aged ≥ 6 years and < 12 years with moderate to severe persistent allergic rhinitis unresponsive to optimal treatment, including daily use of intranasal corticosteroids, will be randomized in a 1:1 ratio to receive FDC desloratadine 0.5mg/mL/prednisolone 4mg/mL - gel for oral administration by Eurofarma Laboratórios SA (experimental drug) or desloratadine 0.5mg/mL - syrup, for five (05) days.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 6 years and ≤ 12 years.
2. Diagnosis of moderate to severe persistent allergic rhinitis (PAR) according to ARIA (Allergic Rhinitis and Its Impact on Asthma) criteria.
3. Sensitization to aeroallergens confirmed by the presence of a positive result on the immediate skin test (PRICK test) and/or by the presence of specific IgE.
4. Total nasal symptom score (TNSS ) ≥ 8 points.
5. Symptom intensity score "nasal obstruction" ≥ 2 points.
6. Signing of the Informed Consent Form (ICF) by the legal guardian and the Informed Assent Form (IAF) before performing any study procedure.

Exclusion Criteria:

1. Being using or having an indication for antibiotic therapy upon selection for the study.
2. Use of prednisolone or other oral corticosteroids in the last seven (07) days.
3. Presence of uncontrolled asthma.
4. Covid-19 diagnosis within four (04) weeks prior to randomization.
5. Positive for SARS-COV-2 rapid antigen test at the time of randomization.
6. Known allergy to desloratadine, prednisolone or any component of the product formulations under investigation.
7. Presence of systemic fungal infections or uncontrolled infections.
8. Presence of any serious or uncontrolled diseases, at the investigator's discretion.
9. Presence of pregnancy or lactation.
10. At the discretion of the investigator, female participants who are already of childbearing age must confirm the use of contraception or expressly declare that they are not at risk of pregnancy because they do not engage in sexual practices or do so in a non-reproductive manner.
11. Participation in a clinical research protocol in the last 6 months, unless, according to the investigator's criteria, their participation in the study could imply a direct benefit for the participant.
12. Presence of any condition that, at the investigator's discretion, renders the patient unfit to participate in the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 262 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-03-23 (Actual); Study Completion 2025-03-23 (Actual)

PRIMARY OUTCOMES:
The total nasal symptom score (TNSS) | five (05) days after the treatment start
  Primary objective: Demonstrate the superiority of the experimental drug (FDC desloratadine 0.5 mg/mL/prednisolone 4 mg/mL from Eurofarma Laboratórios SA) compared to desloratadine 0.5 mg/mL in alleviating symptoms of moderate/severe allergic rhinitis in children through the absolute variation of the total nasal symptom score (TNSS) five (05) days after the treatment start. The TNSS is determined by the sum of the intensity scores attributed to the symptoms of nasal obstruction, runny nose, nasal itching and sneezing in the last 24 hours. Each symptom is assessed using a 4-point categorical scale (0=absent symptom, 1=mild symptom, 2=moderate symptom, 3=intense symptom).

SECONDARY OUTCOMES:
The total nasal symptom score (TNSS) ( efficacy) | three (03) days after the treatment start
  Secondary objectives: To compare the efficacy of the experimental drug (FDC desloratadine 0.5 mg/mL/prednisolone 4 mg/mL from Eurofarma Laboratórios SA) against desloratadine 0.5 mg/mL in alleviating symptoms of moderate/severe allergic rhinitis in children through TNSS. The TNSS is determined by the sum of the intensity scores attributed to the symptoms of nasal obstruction, runny nose, nasal itching and sneezing in the last 24 hours. Each symptom is assessed using a 4-point categorical scale (0=absent symptom, 1=mild symptom, 2=moderate symptom, 3=intense symptom).

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratorios S.A, São Paulo, Brazil